CLINICAL TRIAL: NCT05681715
Title: An Open-label, Crossover Study to Evaluate Rozanolixizumab Self-administration by Study Participants With Generalized Myasthenia Gravis
Brief Title: A Phase 3, Open-label, Crossover Study to Evaluate Self-administration of Rozanolixizumab by Study Participants With Generalized Myasthenia Gravis (gMG)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MG0020; 2022-003870-21 (EudraCT Number)
Record Dates: First submitted 2023-01-04; First posted 2023-01-12 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Generalized Myasthenia Gravis
Keywords: generalized Myasthenia Gravis; gMG; rozanolixizumab
MeSH Terms: conditions — Myasthenia Gravis | interventions — rozanolixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rozanolixizumab Sequence 1: Syringe Driver - Manual Push (Experimental): Study participants will receive predefined weekly doses of rozanolixizumab for 18 weeks.
  Interventions: Drug: Rozanolixizumab
- Rozanolixizumab Sequence 2: Manual Push - Syringe Driver (Experimental): Study participants will receive predefined weekly doses of rozanolixizumab for 18 weeks.
  Interventions: Drug: Rozanolixizumab

INTERVENTIONS:
Drug: Rozanolixizumab — Rozanolixizumab self-administration via Syringe Driver or Manual Push.

SUMMARY:
The purpose of this study is to evaluate the ability of study participants with generalized Myasthenia Gravis (gMG) to successfully self-administer rozanolixizumab after training in the self-administration technique using the syringe driver and manual push methods.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must have a documented diagnosis of generalized Myasthenia Gravis (gMG)
* Study participant is willing to perform and capable of performing home self-administration
* Study participant is considered by the investigator for additional rozanolixizumab treatment with the posology proposed in this study.
* Body weight ≥35 kg
* Study participants may be male or female

Exclusion Criteria:

* Study participant has a known hypersensitivity to other anti-Fc receptor (FcRn) medications, to any components of the study medication, to any of the excipients (including polysorbate 80), or has a known history of hyperprolinemia, since both polysorbate 80 and L-proline are constituents of the rozanolixizumab formulation
* Study participant with a known tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent tuberculosis infection (LTBI), or current or history of nontuberculous mycobacterial infection (NTMBI)
* Study participant has a clinically relevant active infection or a history of serious infection (resulting in hospitalization or requiring IV antibiotic treatment) within 6 weeks before the Baseline Visit
* The study participant previously participated in any rozanolixizumab MG study and met any mandatory withdrawal criteria (unless the reason is directly related to MG0020 participation) or mandatory study drug discontinuation criteria.
* Study participant has received a live vaccination within 4 weeks before starting treatment, or a Bacillus Calmette-Guérin (BCG) vaccine within 1 year before starting treatment; or intends to have a live vaccination during the course of the study or within 8 weeks following the last dose of rozanolixizumab
* Study participant with severe (defined as Grade 3 on the Myasthenia Gravis Activities of Daily Living (MG-ADL) scale) weakness affecting oropharyngeal or respiratory muscles, or who has myasthenic crisis or impending crisis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (27):
- United States (4):
  - Mg0020 50092, Orange, California
  - Mg0020 50099, San Francisco, California
  - Mg0020 50561, Lexington, Kentucky
  - Mg0020 50090, Winston-Salem, North Carolina
- Canada (2):
  - Mg0020 50560, Edmonton
  - Mg0020 50069, Toronto
- Georgia (3):
  - Mg0020 20161, Tbilisi
  - Mg0020 20165, Tbilisi
  - Mg0020 20305, Tbilisi
- Germany (2):
  - Mg0020 40140, Göttingen
  - Mg0020 40177, Münster
- Italy (3):
  - Mg0020 40144, Milan
  - Mg0020 40146, Pavia
  - Mg0020 40150, Roma
- Japan (4):
  - Mg0020 20068, Chiba
  - Mg0020 20078, Hanamaki-shi
  - Mg0020 20077, Sendai
  - Mg0020 20076, Shinjuku-ku
- Poland (3):
  - Mg0020 40155, Gdansk
  - Mg0020 40727, Lodz
  - Mg0020 40153, Poznan
- Mg0020 40729, Niš, Serbia
- Spain (3):
  - Mg0020 40160, Barcelona
  - Mg0020 40267, Barcelona
  - Mg0020 40308, San Sebastián de los Reyes
- United Kingdom (2):
  - Mg0020 40168, Nottingham
  - Mg0020 40163, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- [Result] Bril V, Antozzi C, Berkowicz T, Druzdz A, Gandhi Mehta RK, Mahuwala ZK, Zschuntzsch J, Boehnlein M, Kerbusch V, Lavrov A, Morris M, Singh P, Leite MI. Self-administration of rozanolixizumab via manual push and infusion pump methods in patients with generalised myasthenia gravis: a randomised, phase 3, open-label, crossover study. J Neurol. 2025 Oct 11;272(10):686. doi: 10.1007/s00415-025-13420-6. PMID 41074934

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in April 2023 and concluded in April 2024.
Pre-assignment Details: Participant Flow refers to Safety Set (SS) for Training Period and Randomized Safety Set (RSS) for Self-administration Periods 1 and 2.
Groups:
- All Participants: Training Period: All participants received weekly doses of subcutaneous rozanolixizumab (RLZ) as per their body weight. During the Training Period, the study participants were trained by healthcare professionals on the subcutaneous self-administration of RLZ using both the Syringe Driver (SRD) and Manual Push (MP) methods for 6 weeks before randomization.
- Sequence 1: RLZ Syringe Driver (SRD) - RLZ Manual Push (MP): Randomized participants Self-administered RLZ dose subcutaneously as per their body weight with SRD once every week from Week 7 to 12 during Self-administration Period 1 followed by RLZ administered subcutaneously with MP once every week from Week 13 to 18 during Self-administration Period 2. Study has no wash-out period.
- Sequence 2: RLZ MP - RLZ SRD: Randomized participants Self-administered RLZ dose subcutaneously as per their body weight with MP once every week from Week 7 to 12 during Self-administration Period 1 followed by RLZ administered subcutaneously with SRD once every week from Week 13 to 18 during Self-administration Period 2. Study had no wash-out period.
Period: Training Period (6-weeks)
Arm/Group | All Participants: Training Period | Sequence 1: RLZ Syringe Driver (SRD) - RLZ Manual Push (MP) | Sequence 2: RLZ MP - RLZ SRD
Started | 62 | 0 | 0
Completed | 55 | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Consent withdrawn by participant (not due to AE) | 1 | 0 | 0
Not completed — Not Eligible for SA but continued in study | 3 | 0 | 0
Period: Self-administration Period 1 (6 Weeks)
Arm/Group | All Participants: Training Period | Sequence 1: RLZ Syringe Driver (SRD) - RLZ Manual Push (MP) | Sequence 2: RLZ MP - RLZ SRD
Started | 0 | 28 | 27
Completed | 0 | 23 | 26
Not Completed | 0 | 5 | 1
Not completed — Diagnosis change to amyotrophic lateral sclerosis | 0 | 1 | 0
Not completed — Consent withdrawn by participant (not due to AE) | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Participant became ineligible for SA | 0 | 1 | 0
Not completed — Missed infusion at Visit 13, SA Period1 incomplete | 0 | 2 | 0
Period: Self-administration Period 2 (6 Weeks)
Arm/Group | All Participants: Training Period | Sequence 1: RLZ Syringe Driver (SRD) - RLZ Manual Push (MP) | Sequence 2: RLZ MP - RLZ SRD
Started | 0 | 25 (Two participants missed Visit 13 (Week 12) during Period 1, so were not counted as having completed Period 1. Both participants continued into Period 2.) | 26
Completed | 0 | 25 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refers to the Safety set which included all study participants who received at least 1 dose of investigational medicinal product (IMP) (partial or full).
Arm/Group | All Participants: Training Period
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (15.7)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 45
  65 - <85 years | 17
  >=85 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5
  Black or African American | 1
  White | 55
  Other/Mixed | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Self-administration of Rozanolixizumab (With Correct Use of Syringe Driver and Manual Push, Respectively) During the Self-administration Period at Visit 13 (Week 12)
Description: Successful self-administration was defined by the participant (i) choosing the correct infusion site, (ii) administering SC, and (iii) delivering the intended dose.
Time Frame: Week 12 (last dose of Self-administration Period 1)
Population: The Full Analysis Set (FAS) consisted of all participants who were included in SS, were randomized, and completed both self-administration periods in accordance with the randomization scheme.
Measure: Number; unit: percentage of participants
Groups:
- Period 1: RLZ SRD: Randomized participants Self-administered RLZ dose subcutaneously as per their body weight with SRD once every week from Week 7 to 12 during Self-administration Period 1.
- Period 1: RLZ MP: Randomized participants Self-administered RLZ dose subcutaneously as per their body weight with MP once every week from Week 7 to 12 during Self-administration Period 1.
Arm/Group | Period 1: RLZ SRD | Period 1: RLZ MP
Number analyzed (Participants) | 18 | 23
percentage of participants | 100 | 100

2. Primary Outcome: Percentage of Participants With Successful Self-administration of Rozanolixizumab (With Correct Use of Syringe Driver and Manual Push, Respectively) During the Self-administration Period at Visit 19 (Week 18)
Description: as for outcome 1
Time Frame: Week 18 (last dose of Self-administration Period 2)
Population: FAS consisted of all participants who were included in SS, were randomized, and completed both self-administration periods in accordance with the randomization scheme.
Measure: Number; unit: percentage of participants
Groups:
- Period 2: RLZ SRD: Randomized participants Self-administered RLZ dose subcutaneously as per their body weight with SRD once every week from Week 13 to 18 during Self-administration Period 2.
- Period 2: RLZ MP: Randomized participants Self-administered RLZ dose subcutaneously as per their body weight with MP once every week from Week 13 to 18 during Self-administration Period 2.
Arm/Group | Period 2: RLZ SRD | Period 2: RLZ MP
Number analyzed (Participants) | 23 | 18
percentage of participants | 100 | 100

3. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) After Syringe Driver or Manual Push Self-administration From Visit 2 (Week 1) up to the End of Study Visit (Visit 21 [Week 26])
Description: An Adverse Event (AE) was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE was defined as an AE starting on or after the date of first administration of rozanolixizumab in the study, up to and including 8 weeks (56 days) after the final dose.
Time Frame: From Week 1 up to the End of Study Visit (Week 26)
Population: SS included all study participants who received at least 1 dose of investigational medicinal product (partial or full). The Randomized Safety Set (RSS) consisted of all participants who were included in SS and were randomized. Here, number of participants analyzed included those participants who were evaluable for the outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- RLZ Total: All study participants who received at least 1 dose of RLZ subcutaneously once every week with SRD or MP in Training Period, SA Period 1 and SA Period 2 for 18 weeks.
Arm/Group | Period 1: RLZ SRD | Period 1: RLZ MP | Period 2: RLZ SRD | Period 2: RLZ MP | RLZ Total
Number analyzed (Participants) | 28 | 27 | 26 | 26 | 62
percentage of participants | 35.7 | 29.6 | 26.9 | 38.5 | 75.8

4. Secondary Outcome: Percentage of Participants With Local Site Reactions up to 24 Hours After Each Administration During the Training Period and Self-administration Periods
Description: The local site reactions up to 24 hours after each administration were defined as AEs reported as local site reactions as per case report form within one day after RLZ administration.
Time Frame: Up to 24 hours after each administration during the Training Period (Baseline to Week 6) and Self-administration Periods (Week 7 to Week 18)
Population: SS included all study participants who received at least 1 dose of investigational medicinal product (partial or full). Here, number of participants analyzed included those participants who were evaluable for the outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants: Training Period | Period 1: RLZ SRD | Period 1: RLZ MP | Period 2: RLZ SRD | Period 2: RLZ MP
Number analyzed (Participants) | 62 | 28 | 27 | 26 | 26
percentage of participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With Medication Errors Associated With Adverse Reactions During the 2 Self-administration Periods of the Study
Description: Medication errors were defined as an unintended failure in the drug treatment process that leads to, or has the potential to lead to, harm to the study participant. Medication Errors associated with adverse reactions during the 2 Self-administration Periods were measured.
Time Frame: During the Self-administration Periods (Week 7 to Week 18)
Population: RSS consisted of all participants who were included in SS and were randomized. Here, number of participants analyzed included those participants who were evaluable for the outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Period 1: RLZ SRD | Period 1: RLZ MP | Period 2: RLZ SRD | Period 2: RLZ MP
Number analyzed (Participants) | 28 | 27 | 26 | 26
percentage of participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Week 1 up to the End of Study Visit (Week 26)
Description: TEAEs were reported for SS and RSS. The RLZ Total arm includes data for all 62 participants from the Training Period to the Safety Follow-Up Period including participants who discontinued during the Training Period or were not randomized but continued in the study.
Groups:
- Self-Administration Period 1 and 2: RLZ SRD: Participants in Sequence 1 (from Week 7 to Week 12) and in Sequence 2 (from Week 13 to Week 18) received weekly doses of RLZ subcutaneously using the SRD administration method.
- Self-Administration Period 1 and 2: RLZ MP: Participants in Sequence 2 (from Week 7 to Week 12) and in Sequence 1 (from Week 13 to Week 18) received weekly doses of RLZ subcutaneously using the MP administration method.
Arm/Group | All Participants: Training Period | Self-Administration Period 1 and 2: RLZ SRD | Self-Administration Period 1 and 2: RLZ MP | RLZ Total
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/54 | 0/53 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/62 | 3/54 | 1/53 | 7/62
Other Adverse Events (participants affected / at risk) | 19/62 | 6/54 | 6/53 | 24/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants: Training Period (N=62) | Self-Administration Period 1 and 2: RLZ SRD (N=54) | Self-Administration Period 1 and 2: RLZ MP (N=53) | RLZ Total (N=62)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants: Training Period (N=62) | Self-Administration Period 1 and 2: RLZ SRD (N=54) | Self-Administration Period 1 and 2: RLZ MP (N=53) | RLZ Total (N=62)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 5 (5)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 3 (5) | 6 (10)
COVID-19 (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 7 (7)
Headache (Nervous system disorders) | 12 (21) | 4 (7) | 1 (1) | 13 (29)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT05681715/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT05681715/SAP_001.pdf